CLINICAL TRIAL: NCT06924814
Title: Technology-Based Distractions for Minor Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 80120
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Procedural Anxiety
Keywords: Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care group (Active Comparator): No immersive technology will be assigned to the participant. Participant will use their own distraction method.
  Interventions: Behavioral: Standard of Care
- Immersive Technology grorup (Experimental): Immersive technologies including VR headsets, a bluetooth haptic device (Buddy Guard), a screen and projector (BERT), and a tablets with a game will be randomly assigned to the participants. Each participant will receive one technological intervention.
  Interventions: Behavioral: Immersive technology

INTERVENTIONS:
Behavioral: Standard of Care — Participant is allowed to use what they will use as a distraction tool while they are receiving treatment.
  Arms: Standard of Care group
Behavioral: Immersive technology — Participants will be randomly assigned to one of the following four groups; VR headsets, a bluetooth haptic device (Buddy Guard), a screen and projector (BERT), and a tablets with a game. Participant's anxiety will be assessed and pre- and post-intervention assessments will be completed.
  Arms: Immersive Technology grorup

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset, Augmented Reality Headset) are more effective than the standard of care (i.e., no technology-based distraction) for decreasing anxiety and pain scores in pediatric patients undergoing various minor procedures (i.e lumbar punctures and cardiac catheterization). The anticipated primary outcome will be a reduction of overall cumulative medication and secondary outcomes include but are not limited to: physician satisfaction, discharge time, pain scores, anxiety scores, and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient age between 4-17
* English speaking
* Parental consent/patient assent
* Undergoing minor procedure(s) at LPCH or Stanford Hospital

Exclusion Criteria:

* Patient does not consent
* Legal guardian not present to obtain consent
* Patient with a significant neurological condition or major developmental disability
* Patient experiencing nausea
* Patient with active infection of the face or hand
* A history of severe motion sickness
* A history of visual problems
* A history of seizures caused by flashing light
* Major surgery within the last 48 hours
* Patients who are clinically unstable or require urgent/emergent intervention
* Patient or parental preference for general anesthesia

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of technological interventions on anxiety levels in patients who undergo minor procedures | baseline, immediately after the intervention
  Participants will complete the Visual Analogue Scale for Anxiety (VAS-A), a self-report scale to measure anxiety levels before and after the technological intervention. The scale is a horizontal line from 0 to 10 with an anchor at 0 indicating "no anxiety" and an anchor at 10 indicating "worst possible anxiety".

SECONDARY OUTCOMES:
Evaluate the effectiveness of technological interventions on pain levels in patients whose age is 4-11 years old and undergo minor procedures | baseline, immediately after the intervention
  The FSP-R is a self-report measure of pain intensity displaying six faces representing equal intervals between the scale values from least pain = 0 to most pain = 10
To evaluate pain levels pre- and post-intervention, participants will complete the Numerical Rating Pain Scale (NRPS) for patients 12-17 years old. | baseline, immediately after the intervention
  The NRPS quantifies pain intensity on a scale from 0, being no pain, to 10, being the worst imaginable pain.
To evaluate patient's, clinician's, and caregiver's satisfaction levels | immediately after the intervention
  To analyze the patient's, clinician's, and caregiver's satisfaction levels, the feedback in the satisfaction survey at the end will be evaluated. The purpose of this analysis is to provide qualitative data on which aspects of the technological intervention the patient received mattered the most to the patient, clinician, and caregiver.
To evaluate the patient's affect during the intervention using HRAD | during minor procedure
  HRAD contains 5-item scale assessing participant's affective state; happy, relaxed, anxious, distressed, with a yes/no answer to cooperation.
To evaluate the patient's cooperation during the intervention using the modified Induction Compliance Checklist (mICC) | during minor procedure
  The mICC score will be recorded by the trained research observers during the minor procedure.11 behaviors that are commonly observed preoperatively will be recorded. Perfect compliance (score of 0) was compared to those that lacked cooperation. mICC will be rated at the time of intervention and only requires one RA.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States